CLINICAL TRIAL: NCT01193530
Title: The Use of Light Therapy for Managing Sleep Disturbances in Patients With Advanced Cancer
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Low Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2009-0738; NCI-2012-01793 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2010-08-31; First posted 2010-09-02 (Estimated); Results first posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Advanced Cancers
Keywords: Sleep Disturbances; Depression; Anxiety; Fatigue; Quality of life
MeSH Terms: conditions — Parasomnias; Depression; Anxiety Disorders; Fatigue | interventions — Ultraviolet Therapy; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bright Light Therapy (Experimental): Daily Bright Light Therapy using Bright Light Litebook device for two 14 day periods.
  Interventions: Other: Bright Light Therapy; Behavioral: Questionnaires; Behavioral: Study Diaries; Device: Bright Light Litebook
- Dim Red Light Therapy (Placebo Comparator): Daily Dim Red Light Therapy (placebo) using control Red Light Litebook device for 14 days then proceed to the open label phase and receive daily bright light for 14 days.
  Interventions: Other: Dim Red Light Therapy; Behavioral: Questionnaires; Behavioral: Study Diaries; Device: Red Light Litebook

INTERVENTIONS:
Other: Bright Light Therapy — 30 minutes every day for 14 days. After enrollment on day 0, blinded phase of study intervention (i.e. daily bright light or red light) from day 1 to day 14+/-3, then proceed to the open label phase and receive daily bright light between day 15+/-3 and day 28+/-3.
  Arms: Bright Light Therapy
Other: Dim Red Light Therapy — From day 1 to day 14+/-3, daily dim red light therapy for 30 minutes for 14 days where red light device accounts for placebo of the blinded phase of study intervention, then between day 15+/-3 and day 28+/-3 open label phase with daily bright light.
  Arms: Dim Red Light Therapy
Behavioral: Questionnaires — Weekly
  Other Names: Survey
Behavioral: Study Diaries — Daily logs
  Other Names: journal
Device: Red Light Litebook — Control red light device produced by Litebook identical in appearance and dimensions to the bright light device, with the exception it emits at wavelength 680nm (i.e. red light) and at an intensity of 50 lux.
  Arms: Dim Red Light Therapy
Device: Bright Light Litebook — Bright light device consists of 60 LEDs with spectral emission peak at approximately 464nm and fluorescent phosphors which provide a broader, secondary spectral peak near 564nm. Collectively the emitted light appears white.
  Arms: Bright Light Therapy

SUMMARY:
The goal of this research study is to learn if a type of light therapy can be used to help patients with advanced cancer who are having difficulty sleeping to sleep better.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to one of two groups:

* Group 1 will receive one type of light therapy for 30 minutes every day for 14 days.
* Group 2 will receive a placebo light for 30 minutes every day for 14 days. The placebo light is not designed to have any effect on your sleep.

You will not know which group you are in. After 14 days, both groups will begin receiving the light therapy for another 14 days.

Litebook:

You will use a device called a Litebook to receive either the light therapy or the placebo light for 30 minutes, within 2 hours of waking up every day. The Litebook is about the size of a deck of cards. To use the Litebook, you will place it on a table within 2 feet of you while you are sitting down. The Litebook will either deliver the light therapy or the placebo light. You do not need to look directly into the Litebook and you can do usual activities such as eating or reading while you are using it. The study staff will teach you how to use the Litebook.

Study Diaries:

You will complete the following diaries at the end of each day of the 28-day study period:

* The light exposure diary about how much light you were exposed to.
* The sleep diary about your sleeping habits.

It should take about 5 minutes each day to make entries in the study diaries. You will return the diaries to the study staff at 2 weeks and 4 weeks.

You will also wear a watch that will measure your activity level for 24 hours a day while you are on study. You will return the watch to the study staff after you have completed the study.

Questionnaires:

You will complete a questionnaire about any symptoms you are having from the light therapy at the beginning of the study, at 1 week, at 2 weeks, and at 4 weeks. The questionnaire at 1 week can be done over the phone. It should take about 5 minutes to complete.

You will complete the following questionnaires at the beginning of the study, at 2 weeks, and at 4 weeks:

* The Edmonton Symptom Assessment Scale. You will rate 10 symptoms such as tiredness, shortness of breath, pain, and nausea.
* The FACIT-F questionnaire about how well you are able to perform the normal activities of daily living, your quality of life, and how tired you are.
* The HADS questionnaire about your mood.
* The Pittsburgh Sleep Quality Index about your sleep quality, how long you sleep, and any difficulties you are having when you are trying to sleep.

It should take about 25 minutes to complete all of the questionnaires.

Length of Study:

You will be on study for 28 days.

This is an investigational study. The use of light therapy in patients with difficulty sleeping is investigational. It is currently being used for research purposes only.

Up to 152 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced cancer patients seen in Supportive Care outpatient clinic at M.D. Anderson Cancer Center, with average sleep disturbance >=4 out of 10 for at least one week
2. Age 18 or greater
3. Karnofsky performance status score of >=40 at time of inclusion into study
4. Agrees to return to MD Anderson Cancer Center (MDACC) for follow-up visits
5. English speaking

Exclusion Criteria:

1. Persons with congenital blindness and self-reported acquired blindness (independent of the cause) with no light perception
2. Patients with a history of retinal disease
3. Patients with a current diagnosis of major depression disorder or generalized anxiety disorder
4. Patients who have received light therapy in the past either as part of treatment for other disorders or as a study subject
5. Patients currently on amiodarone, thiazide diuretics or epidermal growth factor receptor (EGFR) inhibitors (erlotinib, gefitinib, cetuximab, panitumumab)
6. Patients who are currently receiving ultraviolet A light/ultraviolet B light (UVA/UVB) therapy or tanning sessions at salons
7. Patients with a diagnosis of obstructive sleep apnea or narcolepsy
8. Patients with >2 hours of direct exposure to outdoor natural light per day (light exposure diary -- screening).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rony Dev, DO, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: June 16, 2011 to February 08, 2012. All recruitment done at The University of Texas MD Anderson.
Pre-assignment Details: Study was halted early due to low accrual, many prospective participants did not meet inclusion and exclusion criteria.
Period: Overall Study
Arm/Group | Bright Light Therapy | Dim Red Light Therapy
Started | 4 | 8
Completed | 1 | 3
Not Completed | 3 | 5
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Began Contraindicated Therapy | 1 | 0
Not completed — Lost Light Box | 0 | 1
Not completed — Returned home - out of state | 0 | 1
Not completed — Non-Compliance | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bright Light Therapy | Dim Red Light Therapy | Total
Number analyzed (Participants) | 4 | 8 | 12
Age, Continuous [Median (Full Range); unit: years] | 53 [37 to 66] | 49 [24 to 77] | 50 [24 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 4 | 8 | 12

OUTCOME MEASURES:

1. Primary Outcome: Effect of Bright Light Therapy on Sleep Disturbances Compared to Dim Red Light in Patients With Advanced Cancer Followed at a Palliative Care Outpatient Clinic at a Comprehensive Cancer Center
Description: Pittsburgh Sleep Quality Index (PSQI) measured at baseline and two weeks. The PSQI is a validated tool for insomnia, an effective instrument for measuring the quality and patterns of sleep using a 19-item questionnaire. It differentiates "poor" from "good" sleep by measuring seven areas: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction over the last month. Each area is rated from 0-3 with the higher score reflecting more severe sleep complaints. The addition of all scores permits the analysis of the participant's overall sleep experience. The PSQI global score ranges from 0 to 21, with a score of 5 or greater indicating significant sleep disturbance.
Time Frame: Baseline and Day 14
Population: Due to low enrollment and participation data was not collected for analysis.
Arm/Group | Bright Light Therapy | Dim Red Light Therapy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 14 days of treatment.
Arm/Group | Bright Light Therapy | Dim Red Light Therapy
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/8
Other Adverse Events (participants affected / at risk) | 3/4 | 6/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bright Light Therapy (N=4) | Dim Red Light Therapy (N=8)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Anxiety (Psychiatric disorders) | 1 (1) | 4 (4)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 3 (3)
Depression (Psychiatric disorders) | 1 (1) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 3 (3) | 6 (6)
Flashing vision (Eye disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 3 (3)
Hot flashes (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3) | 5 (5)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 5 (5)
Ocular/Visual (Other) (Eye disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 3 (3) | 6 (6)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Serum triglyceride increased (Investigations) | 1 (1) | 0 (0)
Skin infection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Vascular Changes (Vascular disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 5 (5)
Watering eyes (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes